CLINICAL TRIAL: NCT06918951
Title: Stereotactic Radiotherapy Versus Palliative Conventional Radiotherapy for Oligoprogressive Metastatic Cancers: A Double-Blind Randomized Phase III Trial
Brief Title: Stereotactic Radiotherapy Versus Palliative Conventional Radiotherapy for Oligoprogressive Metastatic Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STOP-2
Record Dates: First submitted 2025-03-10; First posted 2025-04-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Oligoprogression; Oligometastatic Disease; OligoProgressive Metastatic Disease
Keywords: SABR; Radiotherapy; Quality of life; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: This study is a phase III, multicenter, double-blind, randomized trial. Participants will be randomized in a 1:1 ratio between conventional palliative radiotherapy (Control Arm; Arm 1) vs. SABR (Experimental Arm; Arm 2) to all sites of oligoprogressing disease.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind trial. Participants, enrolling oncologists, and the statistician will be blinded to trial arm assignment. The Coordinating Centre will not be blinded and will maintain a list of trial arm assignments (unblinding master list, in electronic format and accessible to project managers at the Coordinating Centre). Randomization will occur at the Coordinating Centre, and randomization results will be communicated to the clinical trials unit of the participating centre. The trial arm assignment will not be documented at the participating centre. The trials unit staff at the participating centre will then notify the non-enrolling oncologist of the trial arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Palliative Radiotherapy) (Active Comparator)
  Interventions: Radiation: Palliative radiotherapy
- Experimental Arm (SABR) (Experimental)
  Interventions: Radiation: Stereotactic ablative radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy (SABR) — SABR is a safe and effective modality for metastasis-directed therapy, delivering a high dose of radiotherapy to a small target using conformal techniques. Emerging evidence suggests that SABR for oligoprogressive cancer may extend the duration of systemic therapy, and result in improvements in Progression Free Survival (PFS) and Overall Survival (OS) compared to historic controls.
  Arms: Experimental Arm (SABR)
Radiation: Palliative radiotherapy — Radiotherapy will consist of 8 Gy in 1 fraction to all sites of oligoprogression.
  Participants will continue their current systemic therapy (if already on systemic therapy at the time of oligoprogression event) or continue off systemic therapy (if the participant was not on systemic therapy at the time of the oligorecurrence event).
  Arms: Control Arm (Palliative Radiotherapy)

SUMMARY:
STOP-2 is a phase III multi-institutional double-blind randomized trial. 194 participants will be enrolled in this trial. Participants will be randomized in a 1:1 ratio between the Control Arm vs. the Experimental Arm.

Participants, enrolling oncologists, and the statistician will be blinded to trial arm assignment.

In the control arm, radiotherapy will consist of 8 Gy in 1 fraction to all sites of oligoprogression, and the experimental arm will consist of SABR treatment to all sites of oligoprogression.

Primary Objectives

* To assess the impact of SABR, compared to palliative conventional radiotherapy, on Progression-free survival on next line systemic therapy (PFS-NEST), oncologic outcomes, and Quality of Life (QOL) in participants with 1-5 oligoprogressing lesions.
* To assess the feasibility of the clinical trial in terms of accrual and success of double-blinding.

Secondary Objectives

* To evaluate and compare the impact of SABR and palliative radiation therapy on the overall survival (OS), progression free survival (PFS), polymetastatic progression-free survival (PPFS);
* To assess and compare the proportion of participants receiving additional radiation therapy and other metastasis-directed interventions during follow-up between both arms;
* To compare the impact of SABR and palliative radiation therapy on the time to initiation of the next line of systemic therapy;
* To identify and compare the anatomic sites of disease progression between the experimental (SABR) and control (palliative radiation) arms;
* To compare the treatment related toxicity among participants in each arm;
* To evaluate and compare the quality of life among participants in each arm;
* To assess the cost-effectiveness of the experimental arm compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 or older
2. Able to provide informed consent
3. Histologically confirmed solid malignancy (excluding lymphoma or myeloma) with metastatic disease detected on imaging
4. Biopsy of metastasis at some time prior to enrollment is preferred, but not required
5. ECOG performance status 0-2
6. Life expectancy ≥ 6 months
7. Progression meeting RECIST criteria in up to 5 individual lesions. Progression may be defined as:

   1. Progression of an individual metastasis according to RECIST 1.1 criteria (≥ 20% enlargement of the tumour vs. baseline or nadir, taking as reference the smallest diameter seen prior to starting or during systemic therapy, and associated with a 5 mm minimum increase in size) OR
   2. Unambiguous development of a new metastatic lesion at least 5 mm in size OR
   3. Progressive enlargement of a known metastasis on 2 consecutive imaging studies 2-3 months apart with a minimum 5 mm increase in size from baseline.
   4. A progressing primary tumor is eligible as per the criteria above
8. If the participant is on systemic therapy at the time of oligoprogression:

   The most recent systemic therapy agent must have been delivered for a total of at least 3 months, with an initial partial response (PR), complete response (CR) or stable disease (SD) prior to the development of oligoprogressive lesions
9. If the participant is not on systemic therapy at the time of oligoprogression:

   (i.e., "oligorecurrence"(1), however, included as "oligoprogression" for the purpose of this study protocol):
10. There must be PR, CR or SD persisting for at least 3 months prior to the development of oligoprogressive lesions
11. Participants who are not on systemic therapy at the time of oligoprogression must have other site(s) of disease (metastases or primary tumor) that are stable or resolved and have not received definitive treatment (inclusive of surgery, radical doses of radiotherapy including SABR, or ablation) and are not going to receive SABR.
12. All sites of oligoprogression can be safely treated
13. Restaging completed within 12 weeks prior to randomization (see section 5.1)
14. Negative urine pregnancy test for People of Child-Bearing Potential (POCBP) within 4 weeks of radiotherapy start date.

Exclusion Criteria:

1. Serious medical comorbidities precluding radiotherapy. These include ataxia-telangiectasia or scleroderma, Crohn's disease in participants where the gastrointestinal (GI) tract will receive radiotherapy, or ulcerative colitis where the bowel will receive radiotherapy.

   a. For participants with oligoprogressive lesions in the lung or thorax, this includes interstitial lung disease.
2. Substantial overlap with a previously treated radiation volume. Prior radiotherapy in general is allowed, provided that the composite plan meets dose constraints herein. For participants treated with radiation previously, biological effective dose calculations should be used to equate previous doses to the tolerance doses listed in Appendix 1. A tissue recovery factor may be used in these calculations and if so, must be clearly documented, along with elapsed time from previous radiotherapy, and approved by the local principal investigator.
3. Current malignant pleural effusion, malignant ascites, or leptomeningeal disease
4. Inability to treat all sites of oligoprogressive disease
5. Liver metastases requiring placement of fiducial markers for SABR, as this would compromise successful blinding. Liver metastases are eligible if: 1) they are treated at an institution that offers liver SABR without fiducial markers or 2) pre-existing markers such as surgical clips or calcifications would serve as fiducial markers
6. Brain metastasis > 3.5 cm in size or a total volume of brain metastases greater than 30 cc.
7. Clinical or radiologic evidence of spinal cord compression. Participants can be eligible if surgical resection has been performed.
8. Participants with spine instability as judged by a Spinal Instability Neoplastic Score (SINS) of >12.
9. Dominant brain metastasis requiring surgical decompression
10. For participants with liver metastases; moderate/severe liver dysfunction (Child Pugh B or C)
11. Liver metastases located in the "Biliary no fly zone" defined for this trial as common biliary track, cystic duct and distal branches (1 cm) + 5 mm
12. Surgical resection of all oligoprogression metastases (i.e. no lesion available to be treated with SABR)
13. Pregnant or lactating individuals

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2033-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival on Next Line Systemic Therapy (PFS-NEST) | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Time from randomization to progression (RECIST criteria) beyond next line of systemic therapy or death from any cause or date of last follow-up, whichever occurs first. Next line systemic therapy is the first new systemic therapy initiated after documented disease progression
Evaluation of feasibility of the clinical trial in terms of successful accrual | 12 and 24 months
  Accrual will be measured by the number of participants enrolled in the trial within the specified time frame.
Evaluation of feasibility of the clinical trial in terms of success of double-blinding | 6 weeks
  The success of double-blinding will be measured by providing both the participant and oncologist with a blinding questionnaire asking them to select the suspected trial arm assignment (options include palliative arm, SABR arm, or unknown).

SECONDARY OUTCOMES:
Evaluation of OS, PFS, and PPFS | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  To evaluate and compare the impact of SABR and palliative radiation therapy on the overall survival (OS), progression free survival (PFS), polymetastatic progression-free survival (PPFS);
Time to next line systemic therapy | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  To assess and compare the proportion of participants receiving additional radiation therapy and other metastasis-directed interventions during follow-up between both arms;
Comparing the anatomic sites of disease progression | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  A list of anatomical sites at which there are new or progressing lesions will be collected
Evaluation of the treatment related toxicities | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5 for each organ treated (e.g., liver, lung, bone)
Comparing the quality of life among participants in each arm using Functional Assessment of Cancer Therapy: General (FACT-G) | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Quality of life will be assessed with the FACT-G questionnaire. The FACT-G score ranges from 0 to 108, with higher scores indicating a better quality of life.
Comparing the quality of life among participants in each arm using EuroQol 5-Dimension 5-Level (EQ-5D-5L) | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Quality of life will be assessed with the EQ-5D-5L questionnaire. The EQ-5D-5L index score ranges from -0.224 to 1, with higher scores indicating a better quality of life.
Comparing cost-effectiveness of the arms using the resource utilization forms | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Costs associated with each treatment arm will be measured using resource utilization forms.
Comparing cost-effectiveness of the arms using the EQ-5D-5L | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Costs associated with each treatment arm will be measured using EQ-5D-5L
Evaluation of Tumor Response Rate (TRR) using RECIST Criteria | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Tumor response rate will be assessed using RECIST criteria.
Evaluation of Quality of Life (QOL) using European Organization For Research And Treatment Of Cancer (EORTC QLQ-C30) Questionnaire | 3 months, 6 months, 12 months, 15 months, 18 months, 21 months, 24 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Health-related quality of life will be measured using the EORTC QLQ-C30 questionnaire, covering physical functioning, emotional functioning, and symptom scales.
  This questionnaire consists of 30 items, and the score range is 0-100. On this scale, a higher score indicates a higher (better) level of functioning or a higher (worse) level of symptoms, depending on the type of scale.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer - Surrey, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided